CLINICAL TRIAL: NCT02937844
Title: A Safety and Efficacy Study of Autologous Chimeric Switch Receptor Engineered T Cells Redirected to PD-L1 in Patients With Recurrent Glioblastoma Multiforme
Brief Title: Pilot Study of Autologous Chimeric Switch Receptor Modified T Cells in Recurrent Glioblastoma Multiforme
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Sanbo Brain Hospital (Other)
Collaborators: Marino Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SBNK-2016-016-01
Record Dates: First submitted 2016-07-22; First posted 2016-10-19 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2016-10

CONDITIONS: Glioblastoma Multiforme
MeSH Terms: conditions — Glioblastoma | interventions — Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Anti-PD-L1 CSR T cells (Experimental): Patients will receive lymphodepletion chemotherapy consisting of fludarabine and cyclophosphamide, followed by intravenous infusion of autologous anti- PD-L1 CSR T cells. A standard 3+3 escalation approach will be used to obtain the safe dosage of CAR T cells. The tested CAR T cell dosage ranges from 5×10^4 /kg to 1×10^7 /kg.
  Interventions: Biological: Anti-PD-L1 CSR T cells; Drug: Cyclophosphamide; Drug: Fludarabine

INTERVENTIONS:
Biological: Anti-PD-L1 CSR T cells — Prescribed CSR T cells are infused intravenously to patients in a three-day split-dose regimen（day0,10%; day1, 30%; day2, 60%）.
Drug: Cyclophosphamide — 250 mg/m^2, d1-3
Drug: Fludarabine — 25mg/m^2, d1-3

SUMMARY:
CAR T cell immunotherapy has achieved great success in CD19+ B-cell malignancies. Whether this new generation of cell-based immunotherapy can be applied to solid tumors remain to be investigated, partly due to hostile immune-suppressive tumor microenvironment which favors tumor growth but not immune system. Signaling pathway of programmed death 1 (PD-1) and its ligand PD-L1 plays an important role in suppressing immune response against tumors. PD-L1 is over-expressed in 88% of glioblastoma.

We constructed a chimeric switch receptor (CSR) containing the extracellular domain of PD1 fused to the transmembrane and cytoplasmic domain of the costimulatory molecule CD28. CSR modified T cells are able to recognize PD-L1-expressing tumor cells and transduce signals to activate T cells, which results in tumor killing. A truncated EGFR (tEGFR) which lacks of the ligand binding domain and cytoplasmic kinase domain of wildtype EGFR is incorporated into the CSR vector and is used for in vivo tracking and ablation of CSR T cells when necessary. This pilot study is to determine the safety and efficacy of autologous CSR T cells in patients with recurrent glioblastoma.

ELIGIBILITY:
Inclusion Criteria:

1. abilities to understand and the willingness to provide written informed consent;
2. patients are ≥ 18 and ≤ 70 years old;
3. recurrent glioblastoma patients with measurable tumors. Patients have received standard care of medication, such as Gross Total Resection with concurrent Radio-chemotherapy (~54 - 60 Gy, TMZ). Patients must either not be receiving dexamethasone or receiving ≤ 4 mg/day at the time of leukopheresis;
4. Malignant cells are PD-L1 positive confirmed by IHC;
5. karnofsky performance score (KPS) ≥ 60;
6. life expectancy >3 months;
7. satisfactory bone marrow, liver and kidney functions as defined by the following: absolute neutrophile count ≥ 1500/mm^3; hemoglobin > 10 g/dL; platelets > 100000 /mm^3; Bilirubin < 1.5×ULN; alanine aminotransferase (ALT) or aspartate aminotransferase (AST) < 2.5×ULN; creatinine < 1.5×ULN;
8. peripheral blood absolute lymphocyte count must be above 0.8×10^9/L;
9. satisfactory heart functions;
10. patients must be willing to follow the orders of doctors;
11. women of reproductive potential (between 15 and 49 years old) must have a negative pregnancy test within 7 days of study start. Male and female patients of reproductive potential must agree to use birth control during the study and 3 months post study.

Exclusion Criteria:

1. a prior history of gliadel implantation 4 weeks before this study start or antibody based therapies;
2. HIV positive;
3. hepatitis B infection or hepatitis C infection;
4. history of autoimmune disease, or other diseases require long-term administration of steroids or immunosuppressive therapies;
5. history of allergic disease, or allergy to CAR T cells or study product excipients;
6. patients already enrolled in other clinical study;
7. patients, in the opinion of investigators, may not be eligible or not able to comply with the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-07; Primary Completion 2018-07 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Number of Adverse Events related to CSR T cell infusion | 2 years

SECONDARY OUTCOMES:
Treatment Responses Rate | 4 weeks
  Defined as the proportion of patients who achieved complete remission (CR), partial remission (PR), stable disease(SD), or progressive disease (PD).
Overall Survival Rate | 2 years
Progression-free Survival Rate | 6 months

OTHER OUTCOMES:
Persistence of CSR T cells in patients | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Sanbo Brain Hospital Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided